CLINICAL TRIAL: NCT00630006
Title: Genetic Polymorphisms of Interleukin-10 and TNF-α on Outcome of HCV-Related Chronic Liver Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Allocation: Randomized | Model: Factorial | Masking: None
Other Study IDs: KMUH-IRB-950182
Record Dates: First submitted 2008-02-26; First posted 2008-03-06 (Estimated); Last update posted 2008-03-06 (Estimated); Status verified 2007-07

CONDITIONS: Hepatitis C Virus Infection; Chronic Liver Disease
MeSH Terms: conditions — Hepatitis C | interventions — Tumor Necrosis Factor-alpha; Interleukin-10

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Genetic: TNF-alpha and IL-10

SUMMARY:
The prognosis of chronic hepatitis C virus (HCV)infeciton varies from minimal progressive disease to cirrhosis or hepatocellular carcinoma. Host genetic factors contribute to disease severity. It is known that cytokine gene (including tumor necrosis factor-alpha (TNF-alpha) and interleukin-10 (IL-10) polymorphism affect disease prognosis.This study aims to assess the effect of TNF-alpha and IL-10, and their interaction,on prognosis of HCV-related chronic liver disease

ELIGIBILITY:
Inclusion Criteria:

* Anti-HCV-positive patients

Exclusion Criteria:

* Anti-HCV-negative patients

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Dates: Start 2007-01; Study Completion 2008-12 (Estimated)

PRIMARY OUTCOMES:
cytokine gene polymorphism | years

SECONDARY OUTCOMES:
cytokine gene polymorphism on severity of disease | years

CONTACTS AND LOCATIONS:
Overall Officials: Jen-Eing Jeng, M.D., Principal Investigator — Assistant Professor
Locations (1):
- Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City, Kaohsiung, Taiwan